CLINICAL TRIAL: NCT07146620
Title: Effectiveness of Radial Nerve Mobilization Techniques and Their Interfaces for Treating Chronic Epicondylalgia
Brief Title: Effectiveness of Radial Nerve Mobilization for Chronic Epicondylalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Carlos López de Celis, Lecturer Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER: FIS-2021-11
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Tennis Elbow; Physical Therapy Modalities
MeSH Terms: conditions — Tennis Elbow | interventions — Movement; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Treatment protocol based on massage therapy, pressure release of myofascial trigger points, manual mobilization technique (Mulligan), and Diacutaneous Fibrolysis.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The subjects in this group will receive a physical therapy protocol based on massage therapy, pressure release of myofascial trigger points, manual mobilization technique (Mulligan), neurodynamic mobilization, and a real Diacutaneous Fibrolysis (instrument-assisted soft tissue mobilization). The intervention will be administered once per week for four weeks.
  Interventions: Other: Forearm massage; Other: Pressure release for forearm trigger points; Other: Mulligan mobilization with movement technique; Other: Diacutaneous fibrolysis (Real)
- Control Group (Sham Comparator): The subjects in this group will receive a physical therapy protocol based on massage therapy, pressure release of myofascial trigger points, manual mobilization technique (Mulligan), and a Sham Diacutaneous Fibrolysis (instrument-assisted soft tissue mobilization). The intervention will be administered once per week for four weeks.
  Interventions: Other: Forearm massage; Other: Pressure release for forearm trigger points; Other: Mulligan mobilization with movement technique; Other: Radial Nerve Neurodynamic Mobilization; Other: Diacutaneous Fibrolysis (Sham)

INTERVENTIONS:
Other: Forearm massage — A general massage of the forearm will be performed. The physical therapist perform deep, longitudinal strokes. Pressure will be maintained at a level the patient finds comfortable for 3 minutes.
  Other Names: Soft Tissue Mobilization of the Forearm
Other: Pressure release for forearm trigger points — Pressure will be applied to trigger points in the forearm. This will be done in three sets of 30-second applications, with 30 seconds of rest between each.
  Other Names: Trigger point therapy for the forearm; Ischemic compression of forearm trigger point
Other: Mulligan mobilization with movement technique — A lateromedial glide will be performed. The technique will be applied for three sets of 10 repetitions, with 30 seconds of rest between each set.
  Other Names: Mobilization with Movement (MWM)
Other: Radial Nerve Neurodynamic Mobilization — Three sets of 30 nerve glides will be performed at a rhythm of one second of tension followed by one second of rest. There will be 30 seconds of rest between sets.
  Other Names: Radial Nerve Glides
  Arms: Control Group
Other: Diacutaneous fibrolysis (Real) — A real technique of Diacutaneous fibrolysis will be applied to the forearm region for 5 minutes.
  Other Names: Diacutaneous fibrolysis
  Arms: Intervention Group
Other: Diacutaneous Fibrolysis (Sham) — A sham Diacutaneous Fibrolysis technique (skin pinch) will be applied to the forearm region for 5 minutes.
  Arms: Control Group

SUMMARY:
Effectiveness of radial nerve mobilization techniques and their interfaces for treating chronic epicondylalgia

Intervention: This is a randomized controlled clinical trial that will evaluate the effectiveness of adding radial nerve and its interface mobilization techniques to conventional musculoskeletal treatment.

Participants: Patients over 18 years of age with a diagnosis of chronic epicondylalgia and a positive radial nerve neurodynamic test. Those with previous infiltrations, concomitant pathologies, or contraindications will be excluded.

Study Groups:

* Control Group (n=23): Will receive conventional musculoskeletal treatment.
* Intervention Group (n=23): Will receive the same conventional treatment plus mobilization of the radial nerve and its interfaces.

Primary Outcomes:

* Pain (NPRS).
* Pain and functionality (PRTEE).
* Pressure pain threshold (Algometry).
* Pain-free grip strength (Dynamometry).
* Central sensitization (CSI). Assessments will be conducted at baseline, one week after the last treatment, and 3 months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 18 years old.
* Clinical diagnosis of lateral epicondylalgia.
* Chronic epicondylalgia symptoms for at least 3 months.
* Positive radial nerve neurodynamic test
* Signed informed consent form.

Exclusion Criteria:

* Infiltrations for CE within at least 3 months prior to the study.
* Concomitant problems or mobility issues of the upper limb or cervical spine.
* Contraindications specific to Diacutaneous Fibrolysis or neural mobilization.
* Difficulty understanding and signing the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Numeric Pain Rating Scale. Score from 0 to 10. Zero is equivalent to no pain and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
Pain and Functional Disability | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Patient-Rated Tennis Elbow Evaluation. Score from 0 to 100. Higher score indicates more pain and functional disability and zero indicates no pain and disability.
Handgrip | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Grip strength is assessed in kilograms. The value used is the average of three repetitions.
Pressure pain threshold - Elbow | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Pressure pain threshold at the elbow. The lowest intensity of pressure that the subject perceives as pain when applied to the lateral epicondyle is recorded. The value used will be in kilograms per square centimeter.
Pressure pain threshold - short radial extensor | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Pressure pain threshold at the Short radial extensor.The lowest intensity of pressure that the subject perceives as pain when applied to the short radial extensor is used. The value used will be in kilograms per square centimeter.
Pressure pain threshold - Radial nerve | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Pressure pain threshold at the radial nerve. It is used to record the lowest intensity of pressure that the subject perceives as pain when applied to the radial nerve tunnel. The value used will be in kilograms per square centimeter.
Central sensitization syndrome | From enrollment to the end of treatment (4 weeks), and to the end of the study at 16 weeks.
  Central Sensitization Inventory. The questionnaire is scored on a scale from 0 to 100. A score above 40 is considered to indicate central sensitization.
Subjective perception of clinical evolution | From the 4 week to the end of study at 16 weeks
  Global Rating of Change scale. The scale consists of 15 points, ranging from -7 ("Much worse") to +7 ("Much better"). For clinical interpretation, values below "Somewhat better" or "Somewhat worse" are considered clinically unchanged. Values greater than or equal to "Somewhat better" are considered clinically improved, and values greater than "Somewhat worse" are considered clinically worsened.

IPD SHARING:
Plan to Share IPD: No